CLINICAL TRIAL: NCT00845052
Title: Changing Housestaff Culture and Tracking Housestaff Attitudes Regarding Patient Care and Safety
Brief Title: Survey of Housestaff Attitudes Toward Patient Care and Safety
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 0807009889
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Safety Issues; Patient Care
Keywords: Housestaff; Patient Safety; Patient Care; Focus of Study: To assess safety climate amongst housestaff

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- First group of house staff: First group of house staff to be surveyed
- Second group of house staff: Second group of house staff to be surveyed
- Thirst group of house staff: Third group of house staff to be surveyed

SUMMARY:
Background: The occurrence of medical errors and their deleterious effects on quality of care delivered are widely recognized phenomena in healthcare today. This has spurned an aggressive nationwide campaign to improve the quality of care all hospitals throughout the country. Currently, there are numerous reports of quality improvement initiatives across medical centers in the United States. However, a review of the literature failed to identify any publications regarding targeted resident/housestaff involvement in hospital quality improvement and safety related activities.

Purpose: To investigate and track housestaff attitudes on patient care, patient safety, communication and overall quality within the institution.

Objective: To investigate, analyze and publish the results of this prospective study. The information obtained will help us and others understand whether proactive attempts to change housestaff culture can indeed change attitudes towards the better with regards to patient care and safety. It is assumed that improved attitudes ultimately translates into improved care and safety.

Methods: Each residency coordinator in each clinical department will be asked to distribute a survey, which has already been validated for this type of investigation, to each resident in the respective program (see attachment).

The Vice-President of Medical Affairs will provide a cover letter to help with the process. After a week, a reminder will be distributed by the coordinators to each resident asking them to fill out the survey. The surveys will be filled out anonymously. However, each participant will be asked to note their sex, department and year of postgraduate training. This process will be repeated every eight months until June of 2010. The Housestaff Quality council (HQC) has already distributed and collected this survey. The results of those surveys will be used in a retrospective part of this study. The results of (HQC) survey will be used to establish a baseline of the housestaff attitudes at the New York Presbyterian Hospital-Weill Cornell.

Data will be stored on a password protected computer. The Institutional Review Board (IRB), Office of Human Research Protection and Food and Drug Administration and all appropriate federal oversight agencies may have access to those files.

DETAILED DESCRIPTION:
Each residency coordinator in each clinical department will be asked to distribute a survey, which has already been validated for this type of investigation, to each resident in the respective program

ELIGIBILITY:
Inclusion Criteria:

* Members of housestaff working at New York Presbyterian Hospital - Weill Medical College of Cornell University Exclusion Criteria: Not meeting the inclusion criteria

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Housestaff
Sampling Method: Non-Probability Sample
Enrollment: 674 (Actual)
Dates: Start 2008-07; Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Kerr, MD, MBA, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No